CLINICAL TRIAL: NCT06758856
Title: ABC (Additional Betaine and Choline) Study: Effect of Betaine and Choline Intake on Biomarkers of Metabolic Health in Humans
Brief Title: Effect of Betaine and Choline on Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, Clara Cho, Assistant Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 24-03-006
Record Dates: First submitted 2024-12-18; First posted 2025-01-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-08

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: Betaine; Choline; Overweight; Obesity; Metabolism
MeSH Terms: conditions — Obesity; Overweight | interventions — Betaine; Eggs; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Supplements will be double-blinded, which the order of dietary periods will not be revealed to participants until after the study is completed. Care provider, investigator and outcomes assessor who will be involved in collecting study data will not know the supplement assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Daily 3 whole eggs with daily supplement containing 3 g trimethylglycine (Experimental)
  Interventions: Dietary Supplement: Trimethylglycine; Other: Eggs
- Experimental: No eggs with daily supplement containing 3 g trimethylglycine (Experimental)
  Interventions: Dietary Supplement: Trimethylglycine
- Placebo Comparator: No eggs with daily supplement containing 3 g cellulose (Placebo Comparator)
  Interventions: Dietary Supplement: Cellulose

INTERVENTIONS:
Dietary Supplement: Trimethylglycine — Betaine anhydrous from sugar beets
  Arms: Daily 3 whole eggs with daily supplement containing 3 g trimethylglycine; Experimental: No eggs with daily supplement containing 3 g trimethylglycine
Other: Eggs — 3 whole eggs
  Arms: Daily 3 whole eggs with daily supplement containing 3 g trimethylglycine
Dietary Supplement: Cellulose — Cellulose
  Arms: Placebo Comparator: No eggs with daily supplement containing 3 g cellulose

SUMMARY:
The purpose of this research is to determine whether extra betaine and choline influence metabolic health in adults with overweight and obesity.

DETAILED DESCRIPTION:
Betaine (N,N,N-trimethylglycine or also glycine betaine) is a derivative of choline that functions as an organic osmolyte and participates in one-carbon metabolism as a methyl donor. Betaine is naturally found in beets, wheat and spinach and sold as a food supplement without prescription. Choline is recognized as an essential nutrient that is found in various foods including eggs, nuts and beef, with the major form of choline in food found as phosphatidylcholine. In addition to being oxidized to the methyl donor betaine, choline is a precursor of several compounds involved in neurotransmitter synthesis, lipid metabolism and transport as well as the structural integrity and signaling of cell membranes. Previous studies have reported alterations in one-carbon metabolites in response to a single meal containing different forms of choline, with interindividual variability dependent on genetics and gut microbiota composition. This study will extend to longer-term impact of different forms of choline (betaine as oxidized choline and choline provided from food) with a focus on overweight and obesity, which comprise a predominant portion of the population in North America. The objective of this study is to determine the effect of betaine supplementation with or without food-form choline (eggs) on metabolic health in adults with overweight and obesity. A randomized crossover study design will be employed, which men and women of age 18-70 years with BMI 25-35 kg/m2 will participate in a 14-week study consisting of three 4-week dietary periods: 1) daily consumption of 3 grams of betaine supplement with no eggs; 2) daily consumption of 3 grams of betaine supplement with 3 whole eggs; and 3) daily consumption of 3 grams of cellulose supplement with no eggs, in a random order, each dietary period separated by a 1-week washout break. Blood, urine and fecal samples as well as anthropometric measurements will be collected at baseline, then at weeks 4, 9 and 14. The collected biological samples will be used to measure glucose and lipid markers, one-carbon metabolites and profiling of gut microbiota and genotype to determine interindividual differences in metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant of any race or ethnicity between 18-70 years of age (inclusive) at the time of informed consent
* BMI between 25-35 kg/m2
* Non-smoker
* Willing to consume 3 eggs per day for one dietary period of 4 weeks
* Willing to avoid eggs during the rest of the study including washout period breaks except for eggs that are provided
* Willing to fast before the baseline and dietary period lab visits
* Willing to provide a 24-hr prior day food record at the dietary period lab visits
* Willing to provide or collect biological specimen samples at the baseline and dietary period lab visits
* Willing to follow the study protocol including maintaining usual lifestyle during the entire study

Exclusion Criteria:

* Male or female < 18 years or > 70 years of age at the time of consent
* BMI < 25 kg/m2; or BMI > 35 kg/m2
* Pregnant or planning to become pregnant during the course of the study; currently breastfeeding or postpartum < 6 months
* Use of hormone therapy including birth control pills
* Follows a vegan diet
* Current smoker (any form of nicotine, e-cigarettes, etc)
* Use of recreational drugs (may affect metabolic pathway for choline)
* Presence of chronic illnesses, e.g., heart disease, diabetes, cancer, celiac disease, inflammatory bowel disease (Crohn's disease and ulcerative colitis), gastrointestinal liver or kidney diseases or alcoholism
* Diagnosis of trimethylaminuria (genetic disorder affecting choline use in body)
* Use of antibiotics in the last 2 months
* Use of prebiotics, probiotics or dietary fiber (i.e., Metamucil) supplements in the last 2 months
* Have allergies to eggs or any anaphylactic food allergies
* Have a schedule or lifestyle patterns incompatible with the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Lipid panel | Weeks 0, 4, 9 and 14
  Triglyceride, cholesterol and lipoprotein concentrations
Glucose concentrations | Weeks 0, 4, 9 and 14
  Concentrations of glucose as mol units per volume
Insulin concentrations | Weeks 0, 4, 9 and 14
  Concentrations of insulin as international units per volume
Concentrations of glucose metabolism panel | Weeks 0, 4, 9 and 14
  Concentrations of C-peptide, GLP-1 and GIP as mol units per volume
Body mass | Weeks 0, 4, 9 and 14
  Mass on a scale
One-carbon metabolism panel | Weeks 0, 4, 9 and 14
  Choline metabolite concentrations

SECONDARY OUTCOMES:
Gene expression | Weeks 0, 4, 9 and 14
  Global gene expression in isolated immune cells
Inflammatory response in immune cells | Weeks 0, 4, 9 and 14
  Expression of cytokines in immune cells as assessed in response to lipopolysaccharide challenge
Composition of the gut microbiota | Weeks 0, 4, 9 and 14
  Gut microbiota profiles as assessed by sequencing technologies
Characterization of single nucleotide polymoprhisms | Week 0
  Allelic discrimination of variants in enzymes that influence choline metabolites
Liver health panel | Weeks 0, 4, 9 and 14
  ALT, AST, GGT, ALP and bilirubin concentrations
Blood cell counts | Weeks 0, 4, 9 and 14
  Complete counts of white blood cell, red blood cell, hemoglobin, hematocrit and platelet
Blood pressure | Weeks 0, 4, 9 and 14
  Systolic and diastolic blood pressure
Dietary intake | Weeks 0, 4, 9 and 14
  24-hour prior day food record

CONTACTS AND LOCATIONS:
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeisel SH, da Costa KA. Choline: an essential nutrient for public health. Nutr Rev. 2009 Nov;67(11):615-23. doi: 10.1111/j.1753-4887.2009.00246.x. PMID 19906248
- [Background] Wallace TC, Blusztajn JK, Caudill MA, Klatt KC, Natker E, Zeisel SH, Zelman KM. Choline: The Underconsumed and Underappreciated Essential Nutrient. Nutr Today. 2018 Nov-Dec;53(6):240-253. doi: 10.1097/NT.0000000000000302. Epub 2018 Nov 13. PMID 30853718
- [Background] Lever M, Slow S. The clinical significance of betaine, an osmolyte with a key role in methyl group metabolism. Clin Biochem. 2010 Jun;43(9):732-44. doi: 10.1016/j.clinbiochem.2010.03.009. Epub 2010 Mar 25. PMID 20346934
- [Background] Craig SA. Betaine in human nutrition. Am J Clin Nutr. 2004 Sep;80(3):539-49. doi: 10.1093/ajcn/80.3.539. PMID 15321791
- [Background] Cho CE, Taesuwan S, Malysheva OV, Bender E, Tulchinsky NF, Yan J, Sutter JL, Caudill MA. Trimethylamine-N-oxide (TMAO) response to animal source foods varies among healthy young men and is influenced by their gut microbiota composition: A randomized controlled trial. Mol Nutr Food Res. 2017 Jan;61(1). doi: 10.1002/mnfr.201600324. Epub 2016 Aug 3. PMID 27377678
- [Background] Cho CE, Aardema NDJ, Bunnell ML, Larson DP, Aguilar SS, Bergeson JR, Malysheva OV, Caudill MA, Lefevre M. Effect of Choline Forms and Gut Microbiota Composition on Trimethylamine-N-Oxide Response in Healthy Men. Nutrients. 2020 Jul 25;12(8):2220. doi: 10.3390/nu12082220. PMID 32722424